CLINICAL TRIAL: NCT06749301
Title: Repeatability and Reproducibility of the ADC Map in Head and Neck Cancer. Prospective Multicenter Study
Acronym: ADC/SCC oss
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1861/23
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with primary squamous cell carcinoma (SCC) of the hypopharynx, oropharynx, or oral cavity c: Patients over 18 years of age with primary squamous cell carcinoma of the head and neck (hypopharynx, oropharynx or oral cavity, confirmed by histology) will be prospectively enrolled and, according to standard procedures, will have to undergo an MRI examination for diagnostic purposes.

SUMMARY:
Evaluation of the repeatability and reproducibility of ADC maps in both primary and non-primary lesions lymph nodes in patients with head and neck cancer, using an acquisition protocol Standardized DWI

DETAILED DESCRIPTION:
DWI imaging consists of a spin-echo echo-planar sequence (SE-EPI) that will be acquired with 1.5 T or 3 T tomographs according to the equipment of the individual centers involved, setting the acquisition parameters after the administration of any contrast medium.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years;
* primary squamous cell carcinoma (SCC) of the hypopharynx, oropharynx, or oral cavity; confirmed by histology;
* a lesion visible on at least three consecutive DWI images, with a minimum diameter of 2 cm;
* specific written informed consent;

Exclusion Criteria:

* incomplete acquisition of DWI images;
* presence of artifacts that do not allow quantitative analysis of DWI images;
* performance status 2 or more according to Zubrod.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SCC of the head and neck who, according to standard procedures, will have to undergo an MRI examination fordiagnostic purposes.
  Patients must also meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-03-11 (Estimated); Study Completion 2025-03-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the short-term repeatability of ADC maps in both primary and nodal lesions in patients with squamous cell carcinomas (SCC) of the head and neck | 18 months
  A standardized and shared DWI acquisition protocol will be used at a multicenter level. DWI imaging consists of a spin-echo echo-planar (SE-EPI) sequence that will be acquired with 1.5 T or 3 T tomographs, setting the acquisition parameters, after the administration of the contrast medium (if any) (in order to ensure that the second DWI acquisition is performed under the same conditions as the first). The MRI study must include at least one T2-weighted axial sequence, whose images will be used to support the delineation of the lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS National Cancer Institute "regina Elena", Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided